CLINICAL TRIAL: NCT04704557
Title: Cross Therapy Registry - Oedema Post Market Clinical Follow-up of Safety and Patient Outcomes for Subjects Undergoing Peroneal Nerve Stimulation by Geko™. CTR-Oedema-EU
Brief Title: Cross Therapy Registry - Oedema - EU (CTR-Oedema-EU)
Acronym: CTR-Oedema-EU
Status: Terminated | Type: Observational
Why Stopped: Issues withh recruitment
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FSK-REG-001-EU
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Edema Leg
Keywords: Edema Leg

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: geko Neuromuscular Electro Stimulator (NMES) — Neuromuscular Electro Stimulator (NMES)

SUMMARY:
The geko™ Cross Therapy Registry - Oedema - EU (gekoTM CTR - Oedema- EU) study will prospectively and systematically collect clinical data on all device variants used in standard care pathways for edema management allowing for the monitoring of patient outcomes during a follow-up period of up to twelve months.

DETAILED DESCRIPTION:
The geko™ device has a wide range of clinical applications including the post- operative management of oedema.

Although many short-term acute studies have been completed using the device, little clinical data has been collected on the effect of geko™ use in current standard care pathways for oedema management on patient outcomes during follow-up of up to twelve months.

As the manufacturer of the device, Firstkind Limited has an obligation to collect safety and performance data to comply with current regulations (MDR EU 2017/745 Annex XIV, Part B). Consequently, there is a need for an observational study to provide data to demonstrate patient benefit and regulatory compliance.

The geko™ Cross Therapy Registry - Oedema -EU (gekoTM CTR - Oedema - EU) study will prospectively and systematically collect clinical data on all device variants used in standard care pathways for edema management allowing for the monitoring of patient outcomes during a follow-up period of up to twelve months. This study forms part of the overall Post-Market Clinical Follow-up strategy for the device and Post Market Surveillance (PMS) to support device and performance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and able to provide written informed consent.
* Intact healthy skin at the site of gekoTM device application.
* Subjects receiving gekoTM therapy as part of their standard care for oedema reduction.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Use of any concurrent neuro-modulation device.
* Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
* No involuntary movement of the lower leg/foot at the maximum tolerable device setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been identified to receive gekoTM therapy as part of their standard care for oedema reduction.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Safety: AEs and SAEs | One year
  Safety: determine frequency of adverse events (AEs) and serious AEs (SAEs) whether device related or not and compare rate to historic and published data i.e. gekoTM vs standard of care (SC).
Performance | One year
  Performance: determine frequency of Device Deficiencies (DD) and compare rate to historic and published data i.e. gekoTM vs SC.

SECONDARY OUTCOMES:
Summary of routinely collected performance data | One Year
  Summarize routinely tested and collected performance data, such as patient reported outcome measures and compare to historic and published data i.e. gekoTM vs SC.
Summary of Health Economic Impact | One year
  Summarize health economic impact of gekoTM device on patient outcomes in comparison to SC.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tucker A, Maass A, Bain D, Chen LH, Azzam M, Dawson H, Johnston A. Augmentation of venous, arterial and microvascular blood supply in the leg by isometric neuromuscular stimulation via the peroneal nerve. Int J Angiol. 2010 Spring;19(1):e31-7. doi: 10.1055/s-0031-1278361. PMID 22477572
- [Background] Jawad H, Bain DS, Dawson H, Crawford K, Johnston A, Tucker A. The effectiveness of a novel neuromuscular electrostimulation method versus intermittent pneumatic compression in enhancing lower limb blood flow. J Vasc Surg Venous Lymphat Disord. 2014 Apr;2(2):160-5. doi: 10.1016/j.jvsv.2013.10.052. Epub 2014 Jan 28. PMID 26993181
- [Background] Warwick DJ, Shaikh A, Gadola S, Stokes M, Worsley P, Bain D, Tucker AT, Gadola SD. Neuromuscular electrostimulation viathe common peroneal nerve promotes lower limb blood flow in a below-kneecast: A potential for thromboprophylaxis. Bone Joint Res. 2013 Sep 2;2(9):179-85. doi: 10.1302/2046-3758.29.2000176. Print 2013. PMID 23999610
- [Background] Williams KJ, Moore HM, Davies AH. Haemodynamic changes with the use of neuromuscular electrical stimulation compared to intermittent pneumatic compression. Phlebology. 2015 Jun;30(5):365-72. doi: 10.1177/0268355514531255. Epub 2014 Apr 10. PMID 24722790
- [Background] Zhang Q, Styf J, Ekstrom L, Holm AK. Effects of electrical nerve stimulation on force generation, oxygenation and blood volume in muscles of the immobilized human leg. Scand J Clin Lab Invest. 2014 Aug;74(5):369-77. doi: 10.3109/00365513.2014.898323. Epub 2014 Apr 3. PMID 24697619
- [Background] Yilmaz S, Calbiyik M, Yilmaz BK, Aksoy E. Potential role of electrostimulation in augmentation of venous blood flow after total knee replacement: A pilot study. Phlebology. 2016 May;31(4):251-6. doi: 10.1177/0268355515580473. Epub 2015 Apr 6. PMID 25852131
- [Background] Griffin M, Bond D, Nicolaides A. Measurement of blood flow in the deep veins of the lower limb using the geko neuromuscular electro-stimulation device. Int Angiol. 2016 Aug;35(4):406-10. Epub 2016 Mar 2. PMID 26934561
- [Background] Barnes R, Madden LA, Chetter IC. Fibrinolytic effects of peroneal nerve stimulation in patients with lower limb vascular disease. Blood Coagul Fibrinolysis. 2016 Apr;27(3):275-80. doi: 10.1097/MBC.0000000000000409. PMID 26397885
- [Background] Wainwright TW, Burgess LC, Middleton RG. A feasibility randomised controlled trial to evaluate the effectiveness of a novel neuromuscular electro-stimulation device in preventing the formation of oedema following total hip replacement surgery. Heliyon. 2018 Jul 18;4(7):e00697. doi: 10.1016/j.heliyon.2018.e00697. eCollection 2018 Jul. PMID 30094367
- [Background] Mahmood, Ihsan FRCS (T&O); Chandler, Henry MRCS; Kottam, Lucksy PhD; Eardley, William FRCS (T&O); Rangan, Amar FRCS (T&O); Baker, Paul FRCS (T&O) Neuromuscular Electrostimulation Device Reduces Preoperative Edema and Accelerates Readiness for Theater in Patients Requiring Open Reduction Internal Fixation for Acute Ankle Fracture, Techniques in Foot & Ankle Surgery: Decembe 2020 - Volume 19 - Issue 4 - p 215-219 doi: 10.1097/BTF.0000000000000257
- [Background] Jones NJ, Ivins N, Ebdon V, Hagelstein S, Harding KG. Neuromuscular electrostimulation on lower limb wounds. Br J Nurs. 2018 Nov 8;27(20):S16-S21. doi: 10.12968/bjon.2018.27.Sup20.S16. PMID 30418851
- [Background] Harris C, Duong R, Vanderheyden G, Byrnes B, Cattryse R, Orr A, Keast D. Evaluation of a muscle pump-activating device for non-healing venous leg ulcers. Int Wound J. 2017 Dec;14(6):1189-1198. doi: 10.1111/iwj.12784. Epub 2017 Aug 2. PMID 28770561
- [Background] Harris C, Ramage D, Boloorchi A, Vaughan L, Kuilder G, Rakas S. Using a muscle pump activator device to stimulate healing for non-healing lower leg wounds in long-term care residents. Int Wound J. 2019 Feb;16(1):266-274. doi: 10.1111/iwj.13027. Epub 2018 Nov 20. PMID 30460740
- [Background] Pichonnaz C, Bassin JP, Lecureux E, Currat D, Jolles BM. Bioimpedance spectroscopy for swelling evaluation following total knee arthroplasty: a validation study. BMC Musculoskelet Disord. 2015 Apr 25;16:100. doi: 10.1186/s12891-015-0559-5. PMID 25907994
- [Background] Loyd BJ, Kittelson AJ, Forster J, Stackhouse S, Stevens-Lapsley J. Development of a reference chart to monitor postoperative swelling following total knee arthroplasty. Disabil Rehabil. 2020 Jun;42(12):1767-1774. doi: 10.1080/09638288.2018.1534005. Epub 2019 Jan 22. PMID 30668214
- [Background] Loyd BJ, Stackhouse S, Dayton M, Hogan C, Bade M, Stevens-Lapsley J. The relationship between lower extremity swelling, quadriceps strength, and functional performance following total knee arthroplasty. Knee. 2019 Mar;26(2):382-391. doi: 10.1016/j.knee.2019.01.012. Epub 2019 Feb 14. PMID 30772186
- [Background] Virchow, R. (1856).